CLINICAL TRIAL: NCT04053387
Title: A Long-Term, Open-Label, Extension Study to Evaluate the Safety and Efficacy of Tapinarof Cream, 1% for the Treatment of Plaque Psoriasis in Adults
Brief Title: Long Term Extension Study of Tapinarof for Plaque Psoriasis in Adults (3003)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: IQVIA Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMVT-505-3003
Record Dates: First submitted 2019-07-23; First posted 2019-08-12 (Actual); Results first posted 2022-08-08 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2022-08

CONDITIONS: Plaque Psoriasis
Keywords: Tapinarof; plaque psoriasis,; adult; phase 3; topical; open-label; efficacy; safety; psoriasis; long-term; therapeutic aryl hydrocarbon receptor modulating agent
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: Subjects in this study completed treatment with tapinarof or vehicle in 1 of 2 parent Phase 3 pivotal efficacy and safety studies (Study DMVT-505-3001 or Study DMVT-505-3002). The study will consist of up to 40 weeks of tapinarof cream, 1%, and a 4-week safety follow-up period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tapinarof (DMVT-505) Cream Group (Experimental): Subjects who completed 1 of the phase 3 studies evaluating the safety and efficacy of tapinarof had the option to enter this extension study.
  Subjects entering with a PGA ≥ 1 received treatment with tapinarof cream, 1% until they achieve a PGA = 0, at which time treatment was discontinued and subjects were monitored for durability of response (remittive response). If/when disease worsening occurred, as evidenced by a PGA ≥ 2, treatment was re initiated and continued until a PGA = 0 was achieved.
  Subjects entering with a PGA = 0 had treatment discontinued and were monitored for duration of remittive response. If/when disease worsening occurred, as evidenced by a PGA ≥ 2, treatment was re initiated and continued until a PGA = 0 was achieved.
  This treatment and re treatment pattern of use was continued until the end of the study
  Interventions: Drug: tapinarof cream, 1%

INTERVENTIONS:
Drug: tapinarof cream, 1% — Intermittent use of Tapinarof cream, 1%, applied once daily according to PGA score
  Other Names: DMVT-505

SUMMARY:
This is a long-term, open-label, multicenter, study to evaluate the safety and efficacy of topical tapinarof cream, 1% in adults with plaque psoriasis. Subjects in this study completed treatment in 1 of 2 Phase 3 pivotal efficacy and safety studies (Study DMVT-505-3001 or Study DMVT-505-3002). This study will consist of up to 40 weeks of treatment and a 4-week safety follow-up period.

DETAILED DESCRIPTION:
At the completion of the Week-12 visit of the pivotal study (Baseline [Day 1] in this study), all eligible subjects will be offered enrollment in the long-term extension study. Study visits during the treatment period for all subjects will occur every 4 weeks (± 3 days). The total duration of study participation will be approximately 44 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Completed the 12-week treatment period in 1 of the 2 parent studies (Study DMVT-505-3001 or Study DMVT-505-3002);
2. Male and female subjects
3. Females of child bearing potential and male subjects who are engaging in sexual activity that could lead to pregnancy agree to follow the specified contraceptive guidance while on the study, and for at least 4 weeks after the last exposure to study treatment
4. Capable of giving written informed consent

Exclusion Criteria:

1. Used a prohibited concomitant product or procedure to treat psoriasis during parent study
2. Had a serious adverse event (SAE) that was potentially related to treatment or experienced an adverse event (AE) that led to permanent discontinuation of treatment in the parent study
3. History of or ongoing serious illness or medical, physical, or psychiatric condition(s) that, in the Investigator's opinion, may interfere with the subject's completion of the study
4. Known hypersensitivity to tapinarof

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 763 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Butners, Study Director — Dermavant Sciences GmbH
Locations (100):
- United States (81):
  - Dermavant Investigative Site, Birmingham, Alabama
  - Dermavant Investigative Site, Phoenix, Arizona
  - Dermavant Investigative Site, Bryant, Arkansas
  - Dermavant Investigative Site, Fort Smith, Arkansas
  - Dermavant Investigative Site, Fountain Valley, California
  - Dermavant Investigative Site, Fremont, California
  - Dermavant Investigative Site, Fresno, California
  - Dermavant Investigative Site, Los Angeles, California
  - Dermavant Investigative Site, Northridge, California
  - Dermavant Investigative Site, Oceanside, California
  - Dermavant Investigative Site, San Diego, California
  - Dermavant Investigative Site, Santa Ana, California
  - Dermavant Investigative Site, Santa Monica, California
  - Dermavant Investigative Site, Denver, Colorado
  - Dermavant Investigative Site, Cromwell, Connecticut
  - Dermavant Investigative Site, Boca Raton, Florida
  - Dermavant Investigative Site, Boynton Beach, Florida
  - Dermavant Investigative Site, Hialeah, Florida
  - Dermavant Investigative Site, Margate, Florida
  - Dermavant Investigative Site, Miami, Florida
  - Dermavant Investigative Site, Miramar, Florida
  - Dermavant Investigative Site, Boise, Idaho
  - Dermavant Investigative Site, Rolling Meadows, Illinois
  - Dermavant Investigative Site, Evansville, Indiana
  - Dermavant Investigative Site, Indianapolis, Indiana
  - Dermavant Investigative Site, New Albany, Indiana
  - Dermavant Investigative Site, Plainfield, Indiana
  - Dermavant Investigative Site, Overland Park, Kansas
  - Dermavant Investigative Site, Louisville, Kentucky
  - Dermavant Investigative Site, Owensboro, Kentucky
  - Dermavant Investigative Site, Baton Rouge, Louisiana
  - Dermavant Investigative Site, New Orleans, Louisiana
  - Dermavant Investigative Site, Rockville, Maryland
  - Dermavant Investigative Site, Boston, Massachusetts
  - Dermavant Investigative Site, Bay City, Michigan
  - Dermavant Investigative Site, Clarkston, Michigan
  - Dermavant Clinical Site, Detroit, Michigan
  - Dermavant Investigational Site, Detroit, Michigan
  - Dermavant Investigative Site, Fort Gratiot, Michigan
  - Dermavant Investigative Site, Warren, Michigan
  - Dermavant Investigative Site, Fridley, Minnesota
  - Dermavant Investigative Site, Saint Joseph, Missouri
  - Dermavant Investigative Site, Omaha, Nebraska
  - Dermavant Clinical Site, Las Vegas, Nevada
  - Dermavant Investigative Site, Las Vegas, Nevada
  - Dermavant Investigative Site, East Windsor, New Jersey
  - Dermavant Investigative Site, Hackensack, New Jersey
  - Dermavant Investigative Site, Verona, New Jersey
  - Dermavant Clinical Site, Brooklyn, New York
  - Dermavant Investigative Site, Kew Gardens, New York
  - Dermavant Investigative Site, New York, New York
  - Dermavant Investigative Site, Rochester, New York
  - Dermavant Investigative Site, Stony Brook, New York
  - Dermavant Clinical Site, Watertown, New York
  - Dermavant Investigative Site, Cary, North Carolina
  - Dermavant Investigative Site, High Point, North Carolina
  - Dermavant Investigative Site, Wilmington, North Carolina
  - Dermavant Investigative Site, Winston-Salem, North Carolina
  - Dermavant Investigative Site, Beachwood, Ohio
  - Dermavant Investigative Site, Bexley, Ohio
  - Dermavant Investigative Site, Norman, Oklahoma
  - Dermavant Investigate Site, Norman, Oklahoma
  - Dermavant Clinical Site, Gresham, Oregon
  - Dermavant Investigative Site, Portland, Oregon
  - Dermavant Investigative Site, Pittsburgh, Pennsylvania
  - Dermavant Investigative Site, Johnston, Rhode Island
  - Dermavant Investigative Site, Charleston, South Carolina
  - Dermavant Investigative Site, Nashville, Tennessee
  - Dermavant Investigative Site, Arlington, Texas
  - Dermavant Clinical Site, Bellaire, Texas
  - Dermavant Investigative Site, College Station, Texas
  - Dermavant Investigative Site, Dripping Springs, Texas
  - Dermavant Investigative Site, Houston, Texas
  - Dermavant Clinical Site, Houston, Texas
  - Dermavant Investigative Site, Pflugerville, Texas
  - Dermavant Investigative Site, Plano, Texas
  - Dermavant Investigative Site, San Antonio, Texas
  - Dermavant Investigative Site, Webster, Texas
  - Dermavant Investigative Site, West Jordan, Utah
  - Dermavant Investigative Site, Norfolk, Virginia
  - Dermavant Investigative Site, Spokane, Washington
- Canada (19):
  - Dermavant Investigative Site, Edmonton, Alberta
  - Dermavant Investigative Site, Surrey, Bristish Columbia
  - Dermavant Investigative Site, Surrey, British Columbia
  - Dermavant Investigative Site, Ajax, Ontario
  - Dermavant Clinical Site, Burlington, Ontario
  - Dermavant Investigative Site, Cobourg, Ontario
  - Dermavant Investigative Site, Etobicoke, Ontario
  - Dermavant Investigative Site, Hamilton, Ontario
  - Dermavant Clinical Site, Hamilton, Ontario
  - Dermavant Investigative Site, Markham, Ontario
  - Dermavant Clinical Site, Markham, Ontario
  - Dermavant Investigative Site, North Bay, Ontario
  - Dermavant Investigative Site, Oakville, Ontario
  - Dermavant Investigative Site, Ottawa, Ontario
  - Dermavant Investigative Site, Richmond Hill, Ontario
  - Dermavant Investigative Site, Toronto, Ontario
  - Dermavant Investigative Site, Waterloo, Ontario
  - Dermavant Investigative Site, Windsor, Ontario
  - Dermavant Investigative Site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gold LS, Bruno MJ, Lewitt GM, Hebert AA. Characteristics and management of follicular events and contact dermatitis in patients using tapinarof cream for the treatment of atopic dermatitis or plaque psoriasis. J Dermatolog Treat. 2025 Dec;36(1):2517388. doi: 10.1080/09546634.2025.2517388. Epub 2025 Jul 2. PMID 40600584
- [Derived] Desai SR, Stein Gold L, Cameron MC, Golant A, Lewitt GM, Bruno MJ, Martin G, Brown PM, Rubenstein DS, Butners V, Tallman AM. Tapinarof Cream 1% Once Daily for the Treatment of Plaque Psoriasis: Case Photography of Clinical Outcomes from Three Phase 3 Trials. Dermatol Ther (Heidelb). 2023 Oct;13(10):2443-2460. doi: 10.1007/s13555-023-01008-9. Epub 2023 Sep 11. PMID 37697121

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score: Subjects who completed 1 of the phase 3 studies evaluating the safety and efficacy of tapinarof had the option to enter this extension study.
  Subjects entering with a PGA ≥ 1 received treatment with tapinarof cream, 1% until they achieve a PGA = 0, at which time treatment was discontinued and subjects were monitored for durability of response (remittive response). If/when disease worsening occurred, as evidenced by a PGA ≥ 2, treatment was re initiated and continued until a PGA = 0 was achieved.
  Subjects entering with a PGA = 0 had treatment discontinued and were monitored for duration of remittive response. If/when disease worsening occurred, as evidenced by a PGA ≥ 2, treatment was re initiated and continued until a PGA = 0 was achieved.
  This treatment and re treatment pattern of use was continued until the end of the study
Period: Overall Study
Arm/Group | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score
Started | 763
Completed | 531
Not Completed | 232

BASELINE CHARACTERISTICS:
Groups:
- Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score: Subjects who completed 1 of the phase 3 studies evaluating the safety and efficacy of tapinarof had the option to enter this extension study.
  Subjects entering with a PGA ≥ 1 received treatment with tapinarof cream, 1% until they achieved a PGA = 0, at which time treatment was discontinued and subjects were monitored for durability of response (remittive response). If/when disease worsening occurred, as evidenced by a PGA ≥ 2, treatment was re-initiated and continued until a PGA = 0 was achieved.
  Subjects entering with a PGA = 0 had treatment discontinued and were monitored for duration of remittive response. If/when disease worsening occurred, as evidenced by a PGA ≥ 2, treatment was re initiated and continued until a PGA = 0 was achieved.
  This treatment and re treatment pattern of use was continued until the end of the study.
Arm/Group | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score
Number analyzed (Participants) | 763
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (12.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 315
  Male | 448
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 117
  Not Hispanic or Latino | 641
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 51
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 39
  White | 643
  More than one race | 18
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events and Serious Adverse Events
Description: All AEs reported in this extension study were considered as TEAEs except for those AEs ongoing at the end of the pivotal Phase 3 studies but resolved prior to the Visit 1 date for this extension study.
  All SAEs were deemed unrelated to treatment with tapinarof cream, 1%.
Time Frame: Baseline to 44 weeks
Population: Subjects entering with a PGA = 0 had treatment discontinued. Subjects entering with a PGA ≥ 1 received tapinarof until they achieved a PGA = 0 and had treatment discontinued. If/when disease worsening (PGA ≥ 2) occurred treatment was re-initiated and continued until a PGA = 0 was achieved. This treatment and re-treatment pattern of use was continued until the end of the study. The ITT population includes all subjects who signed the informed consent and enrolled in this extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score
Number analyzed (Participants) | 763
Participants
  Adverse Events | 474
  Serious Adverse Events | 19

2. Primary Outcome: Frequency of Adverse Events and Serious Adverse Events
Description: All AEs reported in this extension study were considered as TEAEs except for those AEs ongoing at the end of the pivotal Phase 3 studies but resolved prior to the Visit 1 date for this extension study. Subjects could have reported more than one TEAE.
  All SAEs were deemed unrelated to treatment with tapinarof cream, 1%.
Time Frame: Baseline to 44 weeks
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score
Number analyzed (Participants) | 763
events
  Adverse Events | 1190
  Serious Adverse Events | 21

3. Primary Outcome: Number of Subjects With Clinically Meaningful Changes From Baseline in Clinical Laboratory Values and Vital Signs
Description: The mean chemistry and hematology parameters were assessed for changes and trends over the course of the study. Shifts from Baseline in chemistry and hematology parameters for individual subjects were assessed for clinical relevance. The number of subjects with clinically significant changes from baseline in laboratory values was assessed for clinical relevance.
Time Frame: Baseline to 40 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score: Subjects who completed 1 of the phase 3 studies evaluating the safety and efficacy of tapinarof had the option to enter this extension study.
  Subjects entering with a PGA ≥ 1 received treatment with tapinarof cream, 1% until they achieve a PGA = 0, at which time treatment was discontinued and subjects were monitored for durability of response (remittive response). If/when disease worsening occurred, as evidenced by a PGA ≥ 2, treatment was re initiated and continued until a PGA = 0 was achieved.
  Subjects entering with a PGA = 0 had treatment discontinued and were monitored for duration of remittive response. If/when disease worsening occurred, as evidenced by a PGA ≥ 2, treatment was re initiated and continued until a PGA = 0 was achieved.
  This treatment and re-treatment pattern of use was continued until the end of the study.
Arm/Group | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score
Number analyzed (Participants) | 763
Participants
  Clinically Meaningful changes in hematology | 0
  Clinically meaningful changes in chemistry | 0
  Clinically meaningful changes in urinalysis | 0
  Clinically meaningful changes in pulse rate | 7
  Clinically meaningful changes in systolic blood pressure | 6
  Clinically meaningful changes in diastolic blood pressure | 16

4. Primary Outcome: Remittive Effect of Treatment Success in Pivotal: Median Time to First Worsening (PGA ≥ 2) While Off Therapy for Subjects Who Entered LTE PGA = 0 (Clear)
Description: Subjects who completed 1 of the phase 3 studies evaluating the safety and efficacy of tapinarof had the option to enter this extension study. Subjects entering with a PGA = 0 had treatment discontinued and were monitored for duration of remittive response. If/when disease worsening occurred, as evidenced by a PGA ≥ 2, treatment was re-initiated and continued until a PGA = 0 was achieved. This outcome measure assesses the median time for subjects entering with a PGA = 0 to first worsening (PGA ≥ 2) while off therapy during this extension study.
  The PGA is an assessment of a subject's psoriasis using a static 5-point scale to grade lesions on the clinical characteristics of erythema, scaling, and plaque thickness/elevation. The PGA ranges from 0 to 4, where 0 = clear, 1= almost clear, 2 = mild, 3 = moderate, and 4 = severe.
Time Frame: Baseline to 44 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days from baseline visit
Arm/Group | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score
Number analyzed (Participants) | 79
days from baseline visit | 115 [85.0 to 168.0]

5. Primary Outcome: Complete Disease Clearance During LTE: Number of Subjects Achieving Disease Clearance PGA =0 (Clear) While on Therapy for Subjects Entered LTE PGA ≥ 1 (Almost Clear)
Description: Subjects who completed 1 of the phase 3 studies evaluating the safety and efficacy of tapinarof had the option to enter this extension study. Subjects entering with a PGA ≥ 1 continued treatment with tapinarof until they achieved a PGA = 0, at which time treatment was discontinued and subjects were monitored for remittive response. If/when disease worsening occurred, as evidenced by a PGA ≥ 2, treatment was re-initiated and continued until a PGA = 0 was achieved. This outcome measure assesses the number of subjects who entered the extension study with a PGA ≥ 1 and achieved complete disease clearance (PGA=0) while on therapy during this extension study.
  The PGA is an assessment of a subject's psoriasis using a static 5-point scale to grade lesions on the clinical characteristics of erythema, scaling, and plaque thickness/elevation. The PGA ranges from 0 to 4, where 0 = clear, 1= almost clear, 2 = mild, 3 = moderate, and 4 = severe. Higher PGA scores represent more severe disease.
Time Frame: Baseline to 44 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score
Number analyzed (Participants) | 680
Participants | 233

6. Primary Outcome: Response During LTE: Number of Subjects Achieving PGA =0 or 1 (Clear or Almost Clear) While on Therapy for Subjects Who Entered LTE With PGA ≥ 2 (Mild)
Description: Subjects who completed 1 of the phase 3 studies evaluating the safety and efficacy of tapinarof had the option to enter this extension study. Subjects entering with a PGA ≥ 1 continued treatment with tapinarof until they achieved a PGA = 0, at which time treatment was discontinued and subjects were monitored for remittive response. If/when disease worsening occurred, as evidenced by a PGA ≥ 2, treatment was re-initiated and continued until a PGA = 0 was achieved.
  This outcome measure assesses the number of these subjects who entered the study with a PGA≥ 2 and achieved a PGA of 0 or 1 (clear or almost clear) while on therapy during this extension study.
  The PGA is an assessment of a subject's psoriasis using a static 5-point scale to grade lesions on the clinical characteristics of erythema, scaling, and plaque thickness/elevation. The PGA ranges from 0 to 4, where 0 = clear, 1= almost clear, 2 = mild, 3 = moderate, and 4 = severe. Higher PGA scores represent more severe disease.
Time Frame: Baseline to 44 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score
Number analyzed (Participants) | 519
Participants | 302

7. Primary Outcome: Remittive Effect of Treatment Success: Number of Subjects Experiencing Worsening (PGA ≥ 2) While Off Therapy for Subjects Who Entered LTE With a PGA = 0 (Clear)
Description: Subjects who completed 1 of the phase 3 studies evaluating the safety and efficacy of tapinarof had the option to enter this extension study. Subjects entering with a PGA = 0 had treatment discontinued and were monitored for duration of remittive response. If/when disease worsening occurred, as evidenced by a PGA ≥ 2, treatment was re-initiated and continued until a PGA = 0 was achieved. This treatment and re-treatment pattern of use was continued until the end of the study. This outcome measure assesses the number of these subjects entering the study with a PGA= 0 who experienced worsening (PGA ≥ 2) while off therapy at least once during this extension study.
  The PGA is an assessment of a subject's psoriasis using a static 5-point scale to grade lesions on the clinical characteristics of erythema, scaling, and plaque thickness/elevation. The PGA ranges from 0 to 4, where 0 = clear, 1= almost clear, 2 = mild, 3 = moderate, and 4 = severe.
Time Frame: Baseline to 44 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score
Number analyzed (Participants) | 79
Participants
  Number of subjects entering with PGA=0 who experienced PGA ≥ 2 at least 1 time during the study | 60
  Number of subjects entering with PGA=0 who never experienced PGA ≥ 2 throughout the study | 19

8. Primary Outcome: Change From Baseline in %BSA Affected
Description: Subjects received treatment with tapinarof intermittently guided by disease severity. This outcome measure assesses the change from baseline in %BSA affected in all subjects, including those on and those off therapy.
  BSA affected was estimated by the handprint method, where the full palmar hand of the subject represented approximately 1% of the total BSA. Body regions are assigned specific number of handprints (hp) with percentage [Head and neck = 10% (10 hp), upper extremities = 20% (20 hp), Trunk (including axillae and groin) = 30% (30 hp), lower extremities (including buttocks) = 40% (40 hp)]. The total %BSA involved was estimated = % involvement
Time Frame: Baseline to 40 weeks
Population: Subjects entering with a PGA = 0 had treatment discontinued. Subjects entering with a PGA ≥ 1 received tapinarof until they achieved a PGA = 0 and had treatment discontinued. If/when disease worsening (PGA ≥ 2) occurred treatment was re-initiated and continued until a PGA = 0 was achieved. This treatment and re treatment pattern of use was continued until the end of the study. The ITT population includes all subjects who signed the informed consent and enrolled in this extension study.
Measure: Mean (Standard Deviation); unit: percentage of BSA affected
Arm/Group | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score
Number analyzed (Participants) | 742
percentage of BSA affected | -2.03 (4.848)

9. Primary Outcome: Percent Change From Baseline in %BSA Affected
Description: Subjects received treatment with tapinarof intermittently guided by disease severity. This outcome measure assesses the % change from baseline in %BSA affected in all subjects, including those on and those off therapy.
  BSA affected was estimated by the handprint method, where the full palmar hand of the subject represented approximately 1% of the total BSA. Body regions are assigned specific number of handprints (hp) with percentage [Head and neck = 10% (10 hp), upper extremities = 20% (20 hp), Trunk (including axillae and groin) = 30% (30 hp), lower extremities (including buttocks) = 40% (40 hp)]. The total %BSA involved was estimated = % involvement
Time Frame: Baseline to 40 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score
Number analyzed (Participants) | 665
percentage change | -18.48 (149.908)

10. Primary Outcome: Mean Duration (Days) of Treatment Course
Description: Subjects who completed 1 of the phase 3 studies evaluating the safety and efficacy of tapinarof had the option to enter this extension study. Subjects entering with a PGA ≥ 1 continued tapinarof until they achieved a PGA = 0, at which time treatment was discontinued. If/when disease worsening occurred, as evidenced by a PGA ≥ 2, treatment was re-initiated and continued until a PGA = 0 was achieved.
  Mean duration (days) of treatment episode = time (days) from date of each PGA ≥ 2 (or PGA ≥ 1 for the first episode) to 1 day before each subsequent PGA = 0.
  The PGA is an assessment of a subject's psoriasis using a static 5-point scale to grade lesions on the clinical characteristics of erythema, scaling, and plaque thickness/elevation. The PGA ranges from 0 to 4, where 0 = clear, 1= almost clear, 2 = mild, 3 = moderate, and 4 = severe. Higher PGA scores represent more severe disease.
Time Frame: Baseline to 40 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score
Number analyzed (Participants) | 735
days | 172.9 (102.17)

11. Primary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Score
Description: Subjects received treatment with tapinarof intermittently guided by disease severity. This outcome measure assesses the change from baseline in PASI score in all subjects, including those on and those off therapy.
  The PASI scoring system combines the assessment of lesion severity and extent of affected area into a single score: 0 (no disease) to 72 (maximal disease). The body is divided into 4 areas for scoring (head, arms, trunk, and legs). Each area is assessed for 3 signs: erythema (redness), induration (plaque thickness), and scale. The severity of each sign in each body area is assessed and scored independently using a 5-point scale, where 0=none, 1=slight, 2=mild, 3=moderate, 4=severe. Each area is also assessed for percent of skin involved: 0 = (0%), 1 = (1-<10%), 2 = (10-<30%), 3 = (30-<50%), 4 = (50 -<70%), 5 = (70-<90%), 6 = (90-100%). Overall PASI = the sum of (individual scores x by a weighted factor for each body region).
Time Frame: Baseline to 40 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score
Number analyzed (Participants) | 741
scores on a scale | -1.80 (4.334)

12. Primary Outcome: Percent Change From Baseline in Psoriasis Area and Severity Index (PASI) Score
Description: Subjects received treatment with tapinarof intermittently guided by disease severity. This outcome measure assesses the % change from baseline in PASI score in all subjects, including those on and those off therapy.
  The PASI scoring system combines the assessment of lesion severity and extent of affected area into a single score: 0 (no disease) to 72 (maximal disease). The body is divided into 4 areas for scoring (head, arms, trunk, and legs). Each area is assessed for 3 signs: erythema (redness), induration (plaque thickness), and scale. The severity of each sign in each body area is assessed and scored independently using a 5-point scale, where 0=none, 1=slight, 2=mild, 3=moderate, 4=severe. Each area is also assessed for percent of skin involved: 0 = (0%), 1 = (1-<10%), 2 = (10-<30%), 3 = (30-<50%), 4 = (50 -<70%), 5 = (70-<90%), 6 = (90-100%). Overall PASI = the sum of (individual scores x by a weighted factor for each body region).
Time Frame: Baseline to 40 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score
Number analyzed (Participants) | 663
percentage change | -11.90 (151.684)

13. Primary Outcome: Change From Baseline in Disease Impact on Daily Activities, as Measured by the Dermatology Life Quality Index (DLQI)
Description: Subjects received treatment with tapinarof intermittently guided by disease severity. This outcome measure assesses change from baseline in disease impact on daily activities, as measured by the DLQI, in all subjects including those on and those off therapy.
  The DLQI is a 10-item PRO measure that assesses the extent to which the skin condition has affected the subject's quality of life over the past week, including 6 domains (daily activities, personal relationships, symptoms and feelings, leisure, work/school, and treatment). The total score (0-30) is the sum of 10 questions with each ranging from 0 to 3. The scoring of each question is as follows: Very much= 3, A lot=2, A little = 1, Not at all = 0, Not relevant = 0, Question unanswered = 0.
  DLQI scores range from 0 to 30, with a higher score indicating a more impaired quality of life.
Time Frame: Baseline to 40 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score
Number analyzed (Participants) | 538
scores on a scale | -2.0 (4.31)

14. Primary Outcome: Percent Change From Baseline in Disease Impact on Daily Activities, as Measured by the Dermatology Life Quality Index (DLQI)
Description: Subjects received treatment with tapinarof intermittently guided by disease severity. This outcome measure assesses % change from baseline in disease impact on daily activities, as measured by the DLQI, in all subjects including those on and those off therapy.
  The DLQI is a 10-item PRO measure that assesses the extent to which the skin condition has affected the subject's quality of life over the past week, including 6 domains (daily activities, personal relationships, symptoms and feelings, leisure, work/school, and treatment). The total score (0-30) is the sum of 10 questions with each ranging from 0 to 3. The scoring of each question is as follows: Very much= 3, A lot=2, A little = 1, Not at all = 0, Not relevant = 0, Question unanswered = 0.
Time Frame: Baseline to 40 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score
Number analyzed (Participants) | 420
percentage change | -37.1 (121.35)

ADVERSE EVENTS:
Time Frame: subject duration: 40 weeks of treatment and a 4 week, safety follow up period Overall duration of study: 16 months
Groups:
- Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score: Subjects who completed 1 of the phase 3 studies evaluating the safety and efficacy of tapinarof had the option to enter this extension study.
  Subjects entering with a PGA ≥ 1 received treatment with tapinarof cream, 1% until they achieve a PGA = 0, at which time treatment was discontinued and subjects were monitored for durability of response (remittive response). If/when disease worsening occurred, as evidenced by a PGA ≥ 2, treatment was re initiated and continued until a PGA = 0 was achieved.
  Subjects entering with a PGA = 0 had treatment discontinued and were monitored for duration of remittive response. If/when disease worsening occurred, as evidenced by a PGA ≥ 2, treatment was re initiated and continued until a PGA = 0 was achieved.
  This treatment and re treatment pattern of use was continued until the end of the study.
  All SAEs were deemed unrelated to treatment with tapinarof cream, 1%.
Arm/Group | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score
All-Cause Mortality (participants affected / at risk) | 1/763
Serious Adverse Events (participants affected / at risk) | 19/763
Other Adverse Events (participants affected / at risk) | 204/763
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score (N=763)
Arrhythmia (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Appendicitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Pelvic inflammatory disease (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous or Intermittent Use of Tapinarof (DMVT-505) Cream According to PGA Score (N=763)
Folliculitis (Infections and infestations) | 173
Dermatitis contact (Skin and subcutaneous tissue disorders) | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT04053387/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT04053387/SAP_001.pdf